CLINICAL TRIAL: NCT05042258
Title: Using Dupilumab to Improve Circadian Function, Sleep and Pruritus in Children With Moderate/Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Amy Paller, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-4161
Record Dates: First submitted 2021-07-27; First posted 2021-09-13 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Atopic Dermatitis; Sleep Disturbance
MeSH Terms: conditions — Dermatitis, Atopic; Parasomnias | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dupilumab administration (Experimental): dupilumab administered in weight based dosage for 12 weeks. The drug will be administered once a week during this time through a subcutaneous injection.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — 12 week dupilumab administration
  Other Names: Dupixent

SUMMARY:
Single center, prospective, Open label study of sleep, pruritus and circadian function pre/post 12-weeks of dupilumab treatment in children 6-17 years old

DETAILED DESCRIPTION:
Subjects will complete two overnight sleep studies, before and after using dupilumab for 12 weeks, to assess the effect of dupilumab on sleep disturbance in eczema patients. These overnight visits will include PSG, blood draws, skin sensors, urine collection, tape stripping, and photography. Subjects will be given dupilumab to use for 12 weeks at home before returning for the second sleep study.

ELIGIBILITY:
Inclusion Criteria:

* Participants, 6-17 years old at time of enrollment.
* Moderate to severe chronic AD inadequately controlled by topical treatment, diagnosed according to Hanifin and Rajka criteria by a pediatric dermatologist or allergist.
* AD severity will be determined at baseline with Validated Investigator Global Assessment (vIGA) score of moderate (3) or severe (4).
* Patient assessed or parent-proxy (under 8 years old) PROMIS sleep disturbance T-score ≥60.
* Willing and able to comply with visits and study-related procedures.
* On stable regimens (consistent use 14 days before Day 1 of study enrollment) of inhaled corticosteroids, topical steroids, and antihistamines.

Exclusion Criteria:

* Poorly controlled asthma (Asthma Control Test ≤19).
* Self-reported sleep disturbance on 2 or more nights in the past 7 days due to allergic rhinitis.
* Use of concomitant medication that causes scratching.
* Major medical condition (such as cancer).
* Active condition that could affect sleep, such as obstructive sleep apnea, restless leg syndrome, insomnia, narcolepsy, severe sleep disordered breathing, severe depression, COVID-19, or hives (urticaria).
* Having applied topical steroids within 7 days of first or second PSG (important for biomarkers assessment).
* Use of systemic immunosuppressant within 30 days of first PSG.
* Having showered or used moisturizers within 12 hours of first or second PSG.
* Unable to communicate in English (some PROMIS questionnaires not available in translation).
* Other contraindication to receiving dupilumab (such as history of allergic reaction to dupilumab or any of its components).
* Pregnancy.
* Clinical blindness (circadian disturbing).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
PROMIS (Patient Reported Outcome Measurement Information System) parent-proxy score | 12 weeks
  Improvement from baseline in PROMIS Parent-Proxy sleep disturbance score (short format 8-item) after 12 weeks post dupilumab initiation. The minimum value is "Never" and the maximum value is "Always". Higher scores mean worse outcomes.
PROMIS patient score | 12 weeks
  Improvement from baseline in PROMIS Patient-reported sleep disturbance score (short format 8-item) after 12 weeks post dupilumab initiation (in children ≥ 8 years old). The minimum value is "Never" and the maximum value is "Always". Higher scores mean worse outcomes.
Wake After Sleep Onset | 12 weeks
  Percentage of patients achieving clinically significant improvement in minutes of Wake After Sleep Onset from baseline to Week 12 on inpatient polysomnography (PSG).

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Lurie Children's Hospital/Northwestern University
Locations (1):
- Lurie Children's Hospital/Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No